CLINICAL TRIAL: NCT05648981
Title: Effectiveness of Photobiomodulation Using Diode Laser on the Reversal of Inferior Alveolar Nerve Block Anesthesia in Children: a Randomized Controlled Clinical Trial
Brief Title: Diode Laser on the Reversal of Inferior Alveolar Nerve Block Anesthesia in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Anesthesia_2022
Record Dates: First submitted 2022-11-01; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental)
  Interventions: Other: Inferior Alveolar Nerve Block administration with laser irradiation
- Control group (Active Comparator)
  Interventions: Other: Inferior Alveolar Nerve Block administration

INTERVENTIONS:
Other: Inferior Alveolar Nerve Block administration with laser irradiation — Patients will receive inferior alveolar nerve block local anesthesia followed by laser irradiation after completion of the operative procedure.
  Arms: Test group
Other: Inferior Alveolar Nerve Block administration — Patients will not receive any laser irradiation after administration of inferior alveolar nerve block local anesthesia.
  Arms: Control group

SUMMARY:
Inevitable problems were reported following the injection of local anesthesia in pediatric dental procedures, which can last until the elimination of soft tissue anesthesia.

Purpose of the study: To evaluate the effectiveness of diode laser photobiomodulation therapy on the reversal of soft tissue anesthesia (STA) in children following inferior alveolar nerve block anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of operative dental procedures, requiring inferior alveolar nerve (IANB) anesthesia.
* Healthy patients (physical status ASA I).
* Definitely positive or positive patients on the Frankl behavior scale.
* No reported allergies to LA, epinephrine or sulfites.
* Normal lip sensation before administration of LA

Exclusion Criteria:

* Patients requiring surgical procedures (i.e. extractions).
* Patients who will show excessive fear to the Transcutaneous Electric Nerve Stimulator (TENS) device and provide a false-positive response on inactivated electrode (absence of current) using the Venham scale.
* Patients who will not be trainable in the standardized lip tapping procedure (could not learn to distinguish the anesthetized numb side from the non-anesthetized side).
* Patients who will not achieve profound numbness after initial LA administration, requiring additional anesthesia using SEM scale.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to recovery of normal lip sensation | For two hours after the procedure
  Patients will be asked to rate the lower lip numbness on the anesthetized side in comparison to the contralateral non-anesthetized side as described previously.
  Patients" responses will be recorded every time as "yes" or "no". the number of minutes elapsed from exposure to laser irradiation to the first reported a normal sensation of the lower lip

SECONDARY OUTCOMES:
Assessment of soft tissue injury | 24 hours after the procedure
  A telephone call will be done inquiring on any trauma, injury, swelling or biting marks on the lower lip after 24 h.
  this will be recorded as Yes/no responses

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt